CLINICAL TRIAL: NCT02818504
Title: SEMEiotic Oriented Technology for Individual's CardiOmetabolic Risk Self- assessmeNt and Self-monitoring
Acronym: SEMEOTICONS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istituto di Fisiologia Clinica CNR (Other)
Collaborators: Centre de Recherche en Nutrition Humaine Rhone-Alpe (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None
Other Study IDs: GA 611516
Record Dates: First submitted 2016-05-09; First posted 2016-06-29 (Estimated); Last update posted 2016-11-04 (Estimated); Status verified 2016-11

CONDITIONS: Cardiovascular Risk Factor
Keywords: obesity; dysglycemia; hypercholesterolemia; lifestyle; smoking; physical activity
MeSH Terms: conditions — Obesity; Hypercholesterolemia; Smoking; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Repeatability and reproducibility study (Experimental): Monitoring of system ("Wize MIrror") measurements with changes in environmental conditions (fasting state, light, temperature)
  Interventions: Other: Wize Mirror
- Validation study (Experimental): Longitudinal monitoring of cardiometabolic risk factors through an user---friendly, unobtrusive, personalized system for lifestyle self---management (the "Wize Mirror")
  Interventions: Other: Wize Mirror

INTERVENTIONS:
Other: Wize Mirror — Interactive mirror which integrates contactless sensors and a touch screen interface to derive a semeiotic model of the face with reference to cardiometabolic risk in healthy subjects

SUMMARY:
Cardio-metabolic risk factors include obesity, physical inactivity, smoke, alcohol abuse, high blood lipids or sugar and arterial hypertension. Systems for self-learning and self-monitoring may help people improve and maintain a healthy lifestyle through tailored suggestions about diet, weight control, physical activity, fatigue,stress.

SEMEOTICONS exploits the human face as an indicator of individual's health status and translates signs obtained from the face using contactless sensors into measures and descriptors to be automatically evaluated by a an interactive smart mirror. This "Wize Mirror" extracts descriptors from videos, images and gas concentration signals and integrates them in a virtual model used to compute and trace the evolution of an individual's wellness index. A health diary enables each individual to evaluate and personally relate his/her lifestyle to his/her well-being. Coaching messages are provided, in relation to the evolution of the wellness index and of each descriptor, to provide useful suggestions on correct lifestyle self-monitoring.

The purpose of this study is assess the accuracy of the information derived from the Wize Mirror in expressing the health status of the individual.

The reproducibility and repeatability study will evaluate whether measurements are stable over short time spans and whether they are influenced by meals light and temperature conditions.

To verify whether the Wize Mirror is able to detect variations in physical and emotional health status with appropriate lifestyle changes, the validation study will cross-check measurements from the Wize Mirror against reference clinical tests at enrolment and after 3 months of personalized suggestions for healthy behavior.

Reference tests include

* Physician visit
* Measurement of blood oxygen content and skin end products of sugar metabolism,body composition, energy expenditure, vascular function
* Laboratory profile and exhaled gas composition
* Questionnaires on quality of life and lifestyle (food, sleep, physical activity, smoking, alcohol, stress).

Wize Mirror measures include

* 3D reconstruction of face images for roundness, color, stress and fatigue
* Heart and respiratory rate
* Detection of skin sugar metabolism end-products and of eye lipid deposits
* Small vessel vasodilating ability with local heating The results will allow to assess whether the Wize Mirror is easy to use and helpful for self-monitoring of cardio-metabolic risk.

DETAILED DESCRIPTION:
Cardio--metabolic (CM) risk is a cluster of risk factors indicative of a patient's overall risk for cardiovascular diseases (CVD), the leading cause of morbidity and mortality worldwide and type-2 diabetes. CM risk factors include obesity, physical inactivity, smoke, alcohol abuse, abnormal lipid metabolism, hyper-glycaemia and arterial hypertension.

Educational programs and lifestyle interventions represent effective tools to improve the risk profile but they need time consuming and expensive counselling and supervision of various health professionals . A rational alternative to intensive individual coaching is the use of systems for self-learning and self-monitoring, to help people change and maintain a healthy lifestyle through tailored suggestions about nutrition, weight control, physical activity, fatigue, and stress.

SEMEOTICONS exploits the human face as an indicator of individual's health status and translates signs obtained from the face into measures and descriptors to be automatically evaluated by a computerized application, an interactive smart mirror, which seamlessly integrates contactless sensors, such as 3D optical sensors, a multispectral camera, gas detection sensors, and microphones and a touch-screen interface for user's interactions and output visualization.

This "Wize Mirror" collects data in the form of videos, images and gas concentration signals, and extracts a number of biometric, morphometric, colorimetric, and compositional descriptors that represent individual's facial signs. The integration of such descriptors constitute a virtual model used to compute and trace the evolution of an individual's wellness index. A health diary about this index enables each individual to evaluate and personally relate his/her lifestyle to his/her well-being. Coaching messages are provided, in relation to the evolution of the wellness index and of each descriptor to provide useful suggestions on correct lifestyle self-monitoring.

The purpose of this study is assess the accuracy of the information derived from the Wize Mirror in expressing the health status of an individual.

Arm 1 Reproducibility and repeatability study (to be performed at the French site Lyon only).

The reproducibility and repeatability study will evaluate whether Wize Mirror measurements are influenced by meals, light and temperature conditions in 6 healthy volunteers Data will be acquired during 4 modules corresponding to different use conditions of the mirror

1. - Changes in the fasting state Under artificial lights and at environment temperature (18-20°C), Wize Mirror measurements will be acquired at baseline in the fasting state and at 30, 60 and 120 minutes after a standardized breakfast during three consecutive days.
2. - Changes in light conditions Wize Mirror measurements will be performed at baseline under artificial lights and at environment temperature (18-20°C) then at 30' under artificial lights and at environment temperature (18-20°C) for 3 times consecutively during the same morning with 20 minutes interval between acquisitions.
3. - Changes in temperature conditions Wize Mirror measurements will be performed at baseline under artificial lights and at environment temperature (18-20°C) then at 30' under artificial lights and at temperature increased to 28- 30°C, for 3 times consecutively during the same morning with 20 minutes interval between acquisitions.
4. - Simultaneous changes in light and temperature conditions Wize Mirror measurements will be performed at baseline under artificial lights and at environment temperature (18-20°C) then at 30' under natural lights and at temperature increased to 28- 30°C, in 6 volunteers for 3 times consecutively during the same morning with 20 minutes interval between acquisitions. The visit will last approximately 3 hours. A breakfast will be offered at the end of the visit.

To assess whether measurements are stable over short time spans one of the 6 volunteers will undergo a last visit for the repeatability study in the fasting state. Wize Mirror measurements will be performed at T0 under artificial lights and at environment temperature (18-20°C) for 10 consecutive times with a 30 minutes interval between acquisitions.

During each visit the following Wize Mirror measurements will be performed:

* face morphometry through 3D reconstruction of face images
* colorimetric analysis
* heart rate and respiratory rate
* autofluorescence detection of protein glycation
* skin cholesterol content
* thermal-induced vasodilation by application of warm air at 42°C temperature to the cheek to study microvascular function
* face expression of stress and fatigue through 3D reconstruction of face images
* exhaled gas analysis for ethanol and carbon dioxide

Arm 2 Validation study. The validation study will check data measured from the Wize Mirror against reference clinical tests in 60 healthy volunteers. To verify whether the Wize Mirror is able to detect variations in physical and emotional health status with appropriate lifestyle changes, measurements will be cross-checked at enrolment and after 3 months of personalized suggestions for healthy behavior.

Healthy volunteers will undergo at recruitment the following for user profiling for baseline CM risk

1. Medical history,
2. Physical examination: anthropometric measurements (body height, body weight, waist circumference, hip circumference) and vital signs (heart/respiratory rate, blood pressure)
3. Body composition (lean mass, fatty mass) by air displacement pletysmography
4. Energy expenditure by indirect calorimetry
5. Peripheral venous blood sampling: hemoglobin, creatinine,Total, HDL, LDL cholesterol, triglycerides, gamma glutamyl transferase, aspartate aminotransferase (AST), alanine aminotransferase (ALT), bilirubin, glucose, insulin, HbA1c
6. Skin accumulation of Advanced Glycation End Products (AGEs)
7. Peripheral arterial tonometry for endothelium-dependent vasodilatation
8. Pulse oxymetry for oxygen saturation
9. Exhaled gas sampling
10. Psychological , knowledge and nutritional tests

    1. measures of psychological well being: Life Orientation Test-Revised (LOT-R); General self efficacy scale (GSES)
    2. measures of anxiety, depression: Beck Anxiety Inventory (BAI); Beck Depression Inventory (BDI-II)
    3. measures of quality of life: Perceived Stress Scale (PSS); Short Form (SF)-12 Health Survey; Insomnia Severity Index (ISI) ; World Health Organization (WHO) (Five) Well Being Index
    4. measures of eating and smoking behaviour and physical activity: WHO STEPwise approach to noncommunicable disease risk factor surveillance (STEPS); Audit C Alcohol ; Fagenstrom's test; International Physical Activity Questionnaire (IPAQ) physical activity; Dietary Approaches to Stop Hypertension (DASH) dietary regimen
    5. measure of motivation to change: Motivation to change physical activity, physical activity (MAC2-AF R) ; motivation to change , nutrition (MAC2- AL R)
    6. measures of health literacy: Newest Vital Sign (NVS) Cardio-metabolic risk scores will be calculated to estimate the CM risk profile

    <!-- -->

    1. Heart-SCORE
    2. Fatty-liver-Index (FLI)
    3. Finnish Type 2 Diabetes Risk Score (FINDRISC)
    4. Homeostasis Model Assessment (HOMA) index

Data acquisition to derive computational descriptors for Wize Mirror functioning will include image (still pictures, videos) acquisition in visible light and infrared band before and after thermal stimulation at 42° C and Exhaled gas sampling using the "Wize Sniffer". During each visit the following Wize Mirror measurements will be performed:

* face morphometry through 3D reconstruction of face images
* colorimetric analysis
* heart rate and respiratory rate
* autofluorescence detection of protein glycation
* skin cholesterol content
* thermal-induced vasodilation by application of warm air at 42°C temperature to the cheek to study microvascular function
* face expression of stress and fatigue through 3D reconstruction of face images
* exhaled gas analysis for ethanol and carbon dioxide

Healthy volunteers will then undergo periodically (minimum time interval 2 weeks) face image acquisition, exhaled gas sampling and they will fill through the Wize Mirror screen lifestyle questionnaires till week 12 (end of study). At the end of study visit they will repeat baseline assessments and fill in a questionnaire to evaluate Wize Mirror ease of use and acceptability.

The changes in Wize Mirror measurements obtained at baseline and end of study will be correlated with changes in body weight, waist circumference and Fatty liver index. Relationship with quality of life, or other well-being questionnaire SCORE, standard biochemistry and specific tests will be also assessed.

ELIGIBILITY:
Inclusion Criteria:

* Blood pressure and heart rate measure after 10 minutes lying without treatment: 95 mmHg<Systolic Blood Pressure<160 mmHg; 45 mmHg<Diastolic Blood Pressure<90 mmHg; 40 bpm<Heart rate<100bpm.
* Broad range of CM risk profile
* Undergoing medical examination at the inclusion visit
* Interested and willing to change their lifestyle by decreasing body weight and/or increasing physical fitness and/or improving their well-being following medical advice

Exclusion Criteria:

* History of overt disease, including hypertension, diabetes, dyslipidemia requiring drug treatment
* Clinical or laboratory findings (lipid, glucose,liver and kidney profile, hemoglobin) at the inclusion visit suggesting any pathological condition requiring treatment
* Chronic medical treatment other than contraception
* Declared pregnancy and breastfeeding
* Claustrophobia
* Minor or adult under guardianship
* Prisoner
* Expected poor compliance
* Subject who has exceeded the maximum foreseen compensation for participation in research protocols

Ages: 25 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 78 (Actual)
Dates: Start 2016-07; Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Plumpness index | 3 months
  a geodetic measure of the roundness of the face as proxy for overweight

SECONDARY OUTCOMES:
Change in Heart Systematic COronary Risk Evaluation (SCORE) | 3 months
  changes in HeartSCORE, an estimate of cardiovascular risk
Change in HOMA-insulin resistance (IR) index | 3 months
  changes in HOMA-insulin resistance (IR) index, an estimate of insulin resistance
Change in Fatty Liver Index | 3 months
  changes in Fatty Liver Index, an estimate of hepatic steatosis
Change in FINDRISC score | 3 months
  changes in FINDRISC, an estimate of the risk of developing type 2 diabetes
Change in % skin autofluorescence by MultiSpectral analysis | 3 months
Change in % suborbital skin fat content by MultiSpectral analysis | 3 months
Change in % Thermal reactive skin hyperemia by MultiSpectral analysis | 3 months
Well being index | 3 months
  Computation of the individual's well-being index from integration of descriptors in the semeiotic model of the face through structural model equations
Intraclass Correlation Coefficient of % skin autofluorescence by MultiSpectral analysis for light changes | Day 15
  Evaluation of the reproducibility of the Wize Mirror measurements with natural or artificial light
Intraclass Correlation Coefficient of % skin autofluorescence by MultiSpectral analysis for temperature changes | Day 15
  Evaluation of the reproducibility of the Wize Mirror measurements at ambient temperature of 18-20 °C and 28-30 °C
Intraclass Correlation Coefficient of % suborbital skin fat content by MultiSpectral analysis for light changes | Day 15
  Evaluation of the reproducibility of the Wize Mirror measurements with natural or artificial light
Intraclass Correlation Coefficient of % suborbital skin fat content by MultiSpectral analysis for temperature changes | Day 15
  Evaluation of the reproducibility of the Wize Mirror measurements at ambient temperature of 18-20 °C and 28-30 °C
Intraclass Correlation Coefficient of Thermal reactive skin hyperemia by MultiSpectral analysis for light changes | Day 15
  Evaluation of the reproducibility of the Wize Mirror measurements with natural or artificial light
Intraclass Correlation Coefficient of Thermal reactive skin hyperemia by MultiSpectral analysis for temperature changes | Day 15
  Evaluation of the reproducibility of the Wize Mirror measurements at ambient temperature of 18-20 °C and 28-30 °C
Score in the System Usability Scale | 3 months (end of study visit)
  Assessment of Wize Mirror acceptability by the end users

CONTACTS AND LOCATIONS:
Overall Officials: Maria Aurora Morales, MD, Principal Investigator — Istiuto di Fisiologia Clinica del CNR Pisa
Locations (3):
- Centre de Recherche en Nutrition Humaine, Lyon, France
- Italy (2):
  - Istituto di Fisiologia Clinica del CNR UOS Milano, Milan, Milano
  - Istituto di Fisiologia Clinica del CNR, Pisa

IPD SHARING:
Plan to Share IPD: No